CLINICAL TRIAL: NCT01012141
Title: Pilot Phase II Study of Docetaxel in Combination With a Dietary Phytonutrient in First Line Treatment of Hormone Independent Metastatic Prostate Cancer
Brief Title: Docetaxel With a Phytochemical in Treating Patients With Hormone Independent Metastatic Prostate Cancer
Acronym: PROTAXY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Principal Investigator, Philippe Chollet, Pr, Centre Jean Perrin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU 793
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2009-11

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Phytochemicals; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: phytochemical
Drug: Docetaxel

SUMMARY:
RATIONALE : Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Dietary supplements, such as phytochemicals, may stop or delay the development of prostate cancer.

DETAILED DESCRIPTION:
The purpose of this study is to assess the pathological response rate in metastatic prostate cancer patients treated by : Docetaxel with a phytochemical

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* WHO performance status 0-2
* Life expectancy ≥ 3 months
* Patients receiving androgen-suppressive therapy in the form of chirurgical castration by orchiectomy or pulpectomy,or medical by LHRH agonist or antagonist with or without anti-androgen or all treatment blocking non gonadic testosterone fraction
* Resulting to testosteronemia <0,5 ng/ml
* Histologically confirmed adenocarcinomia of prostate cancer and documented hormone independant metastatic disease - defined by: objective progression with at least one measurable lesion and/or evaluable lesion according to RECIST criteria and /or a rise in PSA level ("rising PSA")
* Total bilirubin ≤ upper limit of normal (ULN).
* AST and ALT ≤ 1.5 times ULN. Alkaline phosphatase ≤ 2.5 times ULN.
* Serum creatinine < 140 µmol/L or creatinine clearance > 60 mL/ min.
* Neutrophil count > 2.109 L-1.
* Platelet count ≥ 100,000/mm3.
* Hemoglobin ≥ 10 g/dL
* Not previous chemotherapy, except Estracyt
* No liver, kidney or heart failure link to treatment
* No malabsorption syndrome or disease significantly affecting gastrointestinal function
* Prior radiotherapies are permetted withing four weeks of the first study treatment and must be < 25 % of the bone marrow, and all adverse events must be resolved
* Prior surgery are permitted.

Exclusion Criteria:

* Age < 18
* History of psychiatric disorders including psychotic disorder, dementia or seizures that would prohibit the understanding, observance and giving of informed consent
* Previous or concomitant other malignancies except basal or squamous cell carcinoma of the skin or other cancer curatively treated with surgery and/or radiotherapy
* Patients should not have symptomatic brain metastasis
* Concurrent severe and/or uncontrolled co-morbid medical condition
* Malabsorption syndrome or disease significantly affecting gastro-intestinal function or major resection of the stomach, proximal small bowel or grade > 2 dysphagia
* Patients with uncontrolled infection
* History of significant neurologic (i.e. peripheral neuropathy grade > 2 using NCI-CTC criteria v3.0)
* Patients should not have received NSAIDs or COX2 inhibitors within the three weeks prior to starting the study
* Treatment with any investigational drug within 30 days prior to registration
* Patients should not have current regimen containing dietary phytonutrients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Response rate as assessed by clinical, biological and paraclinical examination

SECONDARY OUTCOMES:
Safety as assessed by NCI CTCAE v3.0
To assess the best neuroendocine markers between chromogranin A (CgA), neuron-specific enolase (NSE) and serotonin
Time to progression as assessed by RECIST criteria and PSA level
To assess compliance of per os phytonutrient treatment
Geriatric assessment impact on compliance

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Chollet, MD, Study Chair — Centre Jean Perrin
Locations (2):
- France (2):
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Jean Godinot, Reims